CLINICAL TRIAL: NCT04025333
Title: Helping Ethnic Minority in Hong Kong to Quit Smoking by Understanding Their Knowledge, Attitude and Behavior Related to Smoking
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: UW 18-514
Record Dates: First submitted 2019-06-10; First posted 2019-07-18 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Smoking
Keywords: Smoking Cessation
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims at understanding the needs and concerns of the ethnic minority in Hong Kong, including their behavior, attitudes, and experiences related to smoking and smoking cessation. Specifically, how the level of smoking-related knowledge among them differ from the rest of the Hong Kong people, will be explored. In addition, whether Hong Kong smoking policy influenced the smoking pattern of them will be investigated.

DETAILED DESCRIPTION:
Cigarette smoking is the most significant preventable cause of death and disease, causing 6 million deaths annually worldwide. Despite the fact that tobacco use in Hong Kong has been decreased from 23.3% in 1982 to 10.1% in 2017, the remaining 620 600 daily smokers[3] cannot be overlooked or undervalued.

Hong Kong is a predominantly Chinese society, but it has a sizeable South Asian ethnic minority (EM). According to the Census & Statistics Department, the number of ethnic minorities in Hong Kong increased significantly by 70.8% over the past 10 years. Nevertheless, few smoking and health promotion activities and smoking cessation services have been tailor-made for ethnic minorities in Hong Kong. The barrier of supplying smoking cessation service to the ethnic minority group is that their smoking motivation, willingness to quit, obstacles of quit smoking, attitude towards Hong Kong tobacco law and smoking cessation services are not sure. This will be the first research exploring their knowledge, attitude and experience of cigarette smoking.

ELIGIBILITY:
Inclusion Criteria:

* Only smokers with South Asian(Pakistani, Indian, or Nepalese)backgrounds
* Willing to participate
* aged 18 years or above
* able to speak English
* smoke at least one cigarette per day for the past 3 months

Exclusion Criteria:

* Domestic workers, asylum seekers, refugees, or illegal immigrants, individuals with other ethnic backgrounds, i.e., Africans
* Cannot speak English
* poor cognitive state or active psychotic symptoms, i.e. hallucination, illusion and delusion, noted in the medical records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study only focuses on ethnic minorities. Ethnic minorities refer to persons who reported themselves being of non-Chinese ethnicity in the Population Census/By-census.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
The smoking behaviour among ethnic minorities in Hong Kong. | at the baseline
  Participants were asked about:
  1. The reasons started smoking and the reasons keep smoking behaviour.
  2. The cigarette consumption, the type of cigarettes consumed and the smoking area of ethnic minorities.
  3. The number of quit attempts, the motivation to quit smoking, the ways they overcome withdraw symptoms and depression symptoms as well as reasons they failed to quit.
  4. The reason they don't want to quit smoking.
  5. Whether the above items have changed after they moved from their original countries to Hong Kong.
The knowledge of the risk of smoking in ethnic minorities in Hong Kong. | at the baseline
  Participants were asked about their knowledge of the risk of smoking.
Attitudes towards smoking, tobacco control and smoking cessation in ethnic minorities in Hong Kong. | at the baseline
  Participants were asked about
  1. The attitudes towards smoking, tobacco control policy and smoking cessation.
  2. Their family members' and peers' attitude to their smoking behaviour.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The relevant anonymized patient level data, full dataset, technical appendix, and statistical code are available on reasonable request. The approval from the Principal Investigator for the purpose of data use is required.
Time Frame: After the results of the project has been published.
Access Criteria: Request could be sent to Principal Investigator (william3@hku.hk)